CLINICAL TRIAL: NCT01214941
Title: Effect of Itraconazole and Ticlopidine on the Pharmacokinetics and Pharmacodynamics of Oral Tramadol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Klaus T Olkkola, MD, Prof, Turku University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 54/180/2010; 2010-020617-82 (EudraCT Number)
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2010-10

CONDITIONS: Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Ticlopidine; Itraconazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Ticlopidine (Active Comparator)
  Interventions: Drug: Ticlopidine
- Ticlopidine and itraconazole (Active Comparator)
  Interventions: Drug: Ticlopidine and itraconazole

INTERVENTIONS:
Drug: Placebo — The subjects will be given orally placebo twice a day for 5 days prior to the study.
  Arms: Placebo
Drug: Ticlopidine — The subjects will be given orally ticlopidine 250mg twice a day for 5 days prior to the study.
  Arms: Ticlopidine
Drug: Ticlopidine and itraconazole — The subjects will be given orally ticlopidine 250mg twice a day and itraconazole 200mg as a single daily dose for 5 days prior to the study.
  Arms: Ticlopidine and itraconazole

SUMMARY:
Tramadol is an opioid analgesic, which is widely used in the treatment of acute and neuropathic pain. After oral administration, tramadol is rapidly and almost completely absorbed. Tramadol is extensively metabolised by O- and N-demethylation, which are catalysed by the liver CYP-450 enzymes. O-desmethyltramadol is an active metabolite and its formation is catalysed by CYP2D6. The formation of inactive metabolites is catalysed by CYP3A4 and 2B6. This study is aimed to investigate the possible interaction of oral tramadol with itraconazole and ticlopidine, which are inhibitors of CYP3A4 and 2B6. Twelve healthy male or female adult non-smoking volunteers aged 18-40 years with body weights within ±15% of the ideal weight for height are taken into the study. Primary endpoints of the study are plasma concentrations of tramadol and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18-40
* Body weight within ±15% of the ideal weight for height

Exclusion Criteria:

* A previous history of intolerance to the study drugs or to related compounds and additives
* Concomitant drug therapy of any kind for at least 14 days prior to the study
* Existing or recent significant disease
* History of hematological, endocrine, metabolic or gastrointestinal disease, including gut motility disorders
* History of asthma or any kind of drug allergy
* Previous or present alcoholism, drug abuse, psychological or other emotional problems that are likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements
* A positive test result for urine toxicology
* A "yes" answer to any one of the Abuse Questions
* Pregnancy or nursing
* Donation of blood for 4 weeks prior and during the study
* Special diet or life style conditions which would compromise the conditions of the study or interpretation of the results
* Participation in any other studies involving investigational or marketed drug products concomitantly or within one month prior to the entry into this study
* Smoking for one month before the start of the study and during the whole study period
* Any history of coagulation abnormality, also in first degree relatives

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Concentration of tramadol and its metabolites in plasma | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours after administration of tramadol

SECONDARY OUTCOMES:
Metabolites of tramadol in urine | 0-12 and 12-24 hour fractions after administration of tramadol
  Urine will be collected for 24 hours and M1 and M2 metabolites of tramadol are quantified from 0-12h and 12-24h fractions
Serotonin concentrations | 0, 4 and 8 hours after tramadol administration
  Serotonin concentrations will be analyzed with chromatographical methods from the blood samples drawn 0, 4 and 8 hours after tramadol administration
Pharmacodynamic effects | 1, 2, 3, 4, 5, 6, 8, 10, 12 hours after administration of tramadol
  The psychomotor effects of tramadol will be assessed with the measurement of pupil size with Cogan's pupillometer, Maddox wing test and digit symbol substitution test
Analgesia | 1, 2, 3, 4, 5, 6, 8, 10, 12 hours after the administration of tramadol
  The analgesic effect of tramadol will be evaluated using the cold pressor test. Briefly, the subject's hand is immersed into ice-cold water of + 4° C up to the wrist. The subject is told to keep his or her hand in the water and to report when the cold sensation becomes painful. Cold pain threshold is defined as the latency from the immersion of the hand to the subject's first report of pain. Cold pain intensity is assessed at 30 s intervals following immersion of the hand in cold water for up to 60s . A verbal numerical rating scale of 0-100 will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus T Olkkola, MD, PhD, Prof, Principal Investigator — Turku University Hospital and Turku University
Locations (1):
- Department of Anaesthesiology, Intensive Care, Emergency Care and Pain Medicine, Turku University and Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Hagelberg NM, Saarikoski T, Saari TI, Neuvonen M, Neuvonen PJ, Turpeinen M, Scheinin M, Laine K, Olkkola KT. Ticlopidine inhibits both O-demethylation and renal clearance of tramadol, increasing the exposure to it, but itraconazole has no marked effect on the ticlopidine-tramadol interaction. Eur J Clin Pharmacol. 2013 Apr;69(4):867-75. doi: 10.1007/s00228-012-1433-0. Epub 2012 Oct 26. PMID 23099620